CLINICAL TRIAL: NCT01944345
Title: VariLift Lumbar and Cervical Patient Registry
Brief Title: Patient Registry to Observe Outcomes Following Implantation of the VariLift Interbody Fusion Device
Status: Completed | Type: Observational
Sponsor: Wenzel Spine (Industry)
Responsible Party: Sponsor
Other Study IDs: 2012-001, Ver3
Record Dates: First submitted 2013-09-06; First posted 2013-09-17 (Estimated); Results first posted 2016-04-14 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-04

CONDITIONS: Prolapsed Lumbar Disc; Prolapsed Cervical Disc; Intervertebral Disc Degeneration; Spondylolisthesis, Grade 1; Intervertebral Disc Displacement
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis; Lymphoma, Follicular; Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
The registry has been designed as a prospective, observational program for patients undergoing lumbar or cervical fusion using VariLift device with the ultimate goal to aid in the development of strategic treatment pathways and improved patient care. All patients who agree to participate in the registry will sign an informed consent form and subsequently be treated by their surgeon with the VariLift device. Potential treatment procedures include bilateral posterior lumbar interbody fusion (PLIF), unilateral transforaminal lumbar interbody fusion (TLIF), or bilateral anterior lumbar interbody fusion (ALIF) for the lumbar spine, or cervical unilateral or bilateral ACDF procedure. Surgical procedures can be performed in either an inpatient or outpatient facility. It is anticipated that the VariLift devices will improve patient outcomes and lead to the development of treatment pathways to improve patient care.

DETAILED DESCRIPTION:
The registry is design to collect data prospectively on patients undergoing spinal fusion using the VariLift-L, VariLift-A, or VariLift-C device patients will be enrolled in the registry after reviewing the protocol with their health care provider and signing the informed consent. Data will be collected at recommended time points based on the standards of care of the participating sites. The registry will serve as a database in which retrospective analysis and exploratory analysis of specific research questions will be answered.

Follow up visits will be defined by the treating physicians based on their standard practice. Typical clinical follow up schedules for patients undergoing this type of surgery are pre-operative and 12 months post-operative.

ELIGIBILITY:
Inclusion Criteria:

* Patient is undergoing a procedure with unilateral or bilateral placement of VariLift
* This is the first surgery at the index level
* Patient has understood and signed the informed consent
* Patient is skeletally mature

Exclusion Criteria:

* Revision Surgery
* Is a Worker's Compensation Case
* Infection at the operative site
* Sustained trauma with instability
* Sustained fracture of the vertebra at any of the lumbar spinal levels
* Has a primary diagnosis of degenerative or isthmic spondylolisthesis greater than Grade 1
* Physically or mentally compromised (i.e., being currently treated for a psychiatric disorder, senile dementia, Alzheimer's disease, presence of alcohol or drug abuse)
* Has a diagnosed systemic disease that would affect the subject's welfare or overall outcome of the clinical study (i.e., moderate to severe osteoporosis, Paget's disease, renal osteodystrophy, metastasis to vertebrae, adult onset diabetes, active rheumatoid arthritis, etc.)
* Is an immunologically suppressed or receiving steroid in excess of usual doses
* Is obese (as defined by a Body Mass Index (BMI) of > 40 kg/m2 (BMI equals (weight in pounds x 703) / (height in inches x height in inches))
* Has disabling and daily narcotic dependency greater than 18 months
* Has a known malignancy
* Has a known allergy to metal implants

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing spinal fusion using VariLift lumbar or cervical devices must be screened by the investigating surgeon for eligibility into the registry using the primary diagnosis parameters and the inclusion/exclusion criteria. In addition physicians must follow the associated VariLift Instructions for Use.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2013-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warren Neely, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Foundation Surgical Hospital, San Antonio, Texas
  - Methodist Hospital, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
Data will not be shared

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multi-site recruitment with up to 1000 patients to be enrolled for entire study across all hospital or ASC sites.
Groups:
- Registry Patients: Any patients undergoing lumbar or cervical fusion using the VariLift device in an inpatient or outpatient setting.
Period: Overall Study
Arm/Group | Registry Patients
Started | 69
Completed | 69
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Registry Patients
Number analyzed (Participants) | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 25
Age, Continuous [Median (Full Range); unit: years] | 60 [27 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 29
Region of Enrollment [Number; unit: participants]
  United States | 69
BMI < 40kg/m^2 [Number; unit: participants] | 69

OUTCOME MEASURES:

1. Primary Outcome: Change in Oswestry Disability Index (ODI)/Neck Disability Index (NDI) Score Range 0-50
Description: ODI/NDI Score Range: 0-50 0-4 No disability 5-14 Mild disability 15-24 Moderate disability 25-34 Severe disability >34 Complete disability
Time Frame: Pre-operative and Post-operative 12 months post-operative
Population: Combined cervical and lumbar patients: 30 cervical, 39 lumbar. Mean ODI/NDI was calculated for all patients at preop and 12 month.
Measure: Mean (Standard Deviation); unit: Units on a scale 0-50
Arm/Group | Registry Patients
Number analyzed (Participants) | 69
Units on a scale 0-50
  NDI Score Pre-Surgery | 20.07 (9.37)
  NDI Score at 12 Months | 5.61 (8.15)
  ODI Score at Pre-Surgery | 19.27 (5.33)
  ODI Score at 12 Months | 10.41 (7.20)

2. Primary Outcome: Change in VAS Pain
Description: VAS Pain comparison Preoperative vs post-operative of greater than or equal to 6.
  VAS PAIN SEVERITY SCALE ranges from 0-10. A score of zero (0) means 'no pain' and a ten (10) means 'worst imaginable pain'
Time Frame: Pre-operative and Post-operative 12 months
Population: Total subjects: 30 Cervical subjects, 39 Lumbar subjects. VAS PAIN SEVERITY SCALE ranges from 0-10. Zero = no pain, 10 - worst imaginable pain
Measure: Mean (Standard Deviation); unit: Units on a scale 0-10
Arm/Group | Registry Patients
Number analyzed (Participants) | 69
Units on a scale 0-10
  Cervical Preoperative | 3.53 (1.01)
  Cervical Postoperative | 1.03 (0.38)
  Lumbar Preoperative | 5.85 (0.49)
  Lumbar Postoperative | 2.16 (0.25)

3. Secondary Outcome: Radiological Assessment
Description: Determination of fusion assessment, subsidence or migration of the device and confirmed radiographic dated
Time Frame: Post-operative follow up
Population: 26 (of 30) Cervical Patients 30 (of 39) Lumbar Patients
Measure: Number; unit: participants
Arm/Group | Registry Patients
Number analyzed (Participants) | 69
participants
  Cervical Fusion at 12M | 26
  Cervical Subsidence/Migration (>3mm) | 0
  Lumbar Fusion at 12M | 29
  Lumbar Subsidence/Migration (>3mm) | 1

ADVERSE EVENTS:
Time Frame: Preoperative versus 12 months Postoperative
Description: Events were assessed with each follow-up appointment and as reported by participant.
Arm/Group | Registry Patients
Serious Adverse Events (participants affected / at risk) | 0/69
Other Adverse Events (participants affected / at risk) | 22/69
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Registry Patients (N=69)
Other Not Device Related (Social circumstances) | 22 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days